CLINICAL TRIAL: NCT01825187
Title: Prospective Randomized Controlled Trial Comparing Resident Performance and Clinical Outcomes With Two Different Polypropylene Meshes for Laparoscopic Inguinal Hernias
Brief Title: Prospective Trial Comparing Two Different Polypropylene Meshes for Inguinal Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South East Area Health Education Center, Wilmington, NC (Other)
Collaborators: New Hanover Regional Medical Center (Other)
Responsible Party: Principal Investigator, William Hope, Director of Surgical Education/Assistant Professor of Surgery, South East Area Health Education Center, Wilmington, NC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1302-1
Record Dates: First submitted 2013-03-08; First posted 2013-04-05 (Estimated); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group 1 (Active Comparator): Patients in this group will be randomized to receive the ULTRAPRO mesh
  Interventions: Device: ULTRAPRO Mesh
- Treatment Group 2 (Active Comparator): Patients in this group will be randomized to receive the 3DMAX Mesh
  Interventions: Device: 3DMAX
- Evaluation of Surgical Residents (Other): Surgical residents will be evaluated on the ease of use and the amount of time it takes for them to perform the surgery using these two different meshes.
  Interventions: Other: Evaluation

INTERVENTIONS:
Device: ULTRAPRO Mesh — Patients who are randomized to this group will received ULTRAPRO Mesh for their hernia repair
  Arms: Treatment Group 1
Device: 3DMAX — Patients who are randomized to this group will receive 3DMAX mesh for their hernia repair
  Arms: Treatment Group 2
Other: Evaluation — To evaluate the ease of use and time it takes residents to place and perform the surgery using these two different meshes.
  Arms: Evaluation of Surgical Residents

SUMMARY:
The purpose of this research study is to measure the clinical effectiveness of two different polypropylene meshes used for laparoscopic inguinal hernias by evaluating subjects' length of hospital stay, perioperative complications, recurrence rate, pain score, comfort level and postoperative quality of life. A secondary goal of the study is to evaluate the ease of use and time it takes surgical residents to place the mesh and perform the surgery using these two different meshes.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most common operations performed by general surgeons in the world. There are two main ways to repair an inguinal hernia, open or laparoscopic. Open compared to laparoscopic, is more invasive and leads to more scarring and longer recovery periods. Laparoscopic repair is done by making a small cut in or just below the umbilicus and has become an accepted standard for inguinal hernia repair and has become the technique of choice for recurrent inguinal hernias.

During laparoscopic repair, the placement of a prosthetic mesh aids in reinforcing the abdominal wall and allowing for tension free repair. Meshes also helps to lower the recurrence rate. The most safe and effective type of mesh prosthesis currently being used in laparoscopic inguinal hernia repairs are polypropylene meshes. There is some emerging evidence that "lighter weight" forms of polypropylene meshes may improve quality of life outcomes following surgery for inguinal hernias. Further evaluation is needed to support this evidence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing laparoscopic repair for the treatment of either single or bilateral inguinal hernias
* All surgical residents at New Hanover Regional Medical Center

Exclusion Criteria:

* Subjects requiring emergency surgery
* Pregnant subjects
* Subjects under the age of 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Hope, MD, Principal Investigator — South East Area Health Education Center
Locations (1):
- New Hanover Regional Medical Center, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilezikian JA, Tenzel PL, Johnson RG, Powers WF 4th, Hope WW. A preliminary evaluation of two different meshes in minimally invasive inguinal hernia surgery. Surg Endosc. 2021 Mar;35(3):1342-1347. doi: 10.1007/s00464-020-07512-9. Epub 2020 Mar 30. PMID 32232645

RESULTS

PARTICIPANT FLOW:
Groups:
- ULTRAPRO Mesh Group: Patients in this group will be randomized to receive the ULTRAPRO mesh
  ULTRAPRO Mesh: Patients who are randomized to this group will received ULTRAPRO Mesh for their hernia repair
- 3DMAX Mesh Group: Patients in this group will be randomized to receive the 3DMAX Mesh
  3DMAX: Patients who are randomized to this group will receive 3DMAX mesh for their hernia repair
Period: Overall Study
Arm/Group | ULTRAPRO Mesh Group | 3DMAX Mesh Group | Evaluation of Surgical Residents
Started | 25 | 25 | 25
Completed | 24 | 24 | 24
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: No Baseline Measure data was collected from any Surgical Residents
Groups:
- ULTRAPRO Mesh: Patients in this group will be randomized to receive the ULTRAPRO mesh
  ULTRAPRO Mesh: Patients who are randomized to this group will received ULTRAPRO Mesh for their hernia repair
- 3DMAX Mesh: Patients in this group will be randomized to receive the 3DMAX Mesh
  3DMAX: Patients who are randomized to this group will receive 3DMAX mesh for their hernia repair
- Total: Total of all reporting groups
Arm/Group | ULTRAPRO Mesh | 3DMAX Mesh | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 62 [37 to 87] | 59 [30 to 86] | 61 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 23 | 27
  White | 21 | 1 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Inguinal Hernia Mesh Insertion Times
Description: The primary outcome measure was a comparison of mesh insertion times and were tested using a 2 × 2 ANOVA on the ranked times. Timing of the mesh placement was documented, which included time from mesh insertion in the trocar until completion of mesh fixation. Laparoscopic fixation was performed by placing four tacks; two in the pubic bone, one medial, and one lateral on the upper portion of the mesh. The types of tacks used were AbsorbaTack™ (Medtronics), sutures, CapSure™ (CR Bard) and OptiFix™ (CR Bard). Timing of mesh placement in robotic repairs included mesh placement and the time to place three suture fixation points; one at the pubis, one at the anterior, and 1 at the lateral abdominal wall at the top of the mesh.
Time Frame: During the procedure an average of an hour
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- ULTRAPRO Mesh: ULTRAPRO Mesh: Patients randomized to this group received ULTRAPRO Mesh for their hernia repair
- 3DMAX Mesh: 3DMAX: Patients randomized to this group received 3DMAX mesh for their hernia repair
Arm/Group | ULTRAPRO Mesh | 3DMAX Mesh
Number analyzed (Participants) | 24 | 24
Minutes | 9.76 (7.24) | 8.70 (5.86)
Statistical Analysis 1: Comparison: ULTRAPRO Mesh vs 3DMAX Mesh; Test type: Superiority; p = 0.523, t-test, 1 sided

2. Secondary Outcome: NASA TLX Survey Index Scores
Description: Following surgery, the Hart and Staveland's NASA Task Load Index (TLX) survey was completed by the surgeon to evaluate the surgeon's perceived difficulty and success of the operation. Scale ranges from very low (0) to very high (20) on a 20 point scale (0-20 points). For all outcome measures except performance, 0 indicates the worst outcome and 20 indicates the best outcome. For performance, 0 indicates perfect and 20 indicates failure.
Time Frame: During procedure an average of 1 hour
Measure: Mean (Standard Deviation); unit: Score on NASA scale
Groups:
- ULTRAPRO Mesh Group: NASA TLX Surveys were completed by residents who performed hernia repairs for the arm of subjects who received the UltraPro Mesh.
- 3DMAX Mesh Group: NASA TLX Surveys were completed by residents who performed hernia repairs for the arm of subjects who received the 3DMax Mesh.
Arm/Group | ULTRAPRO Mesh Group | 3DMAX Mesh Group
Number analyzed (Participants) | 24 | 24
Score on NASA scale
  NASA Mental Demand | 7.63 (5.07) | 8.67 (4.20)
  NASA Physical Demand | 6.67 (5.39) | 7.00 (3.88)
  NASA Temporal Demand | 7.46 (4.95) | 8.00 (4.02)
  NASA Performance | 8.04 (5.34) | 6.54 (3.48)
Statistical Analysis 1: Comparison: ULTRAPRO Mesh Group vs 3DMAX Mesh Group; Nasa Mental Demand; Test type: Superiority; p = 0.371, t-test, 1 sided
Statistical Analysis 2: Comparison: ULTRAPRO Mesh Group vs 3DMAX Mesh Group; NASA Physical Demand; Test type: Superiority; p = 0.122, t-test, 1 sided
Statistical Analysis 3: Comparison: ULTRAPRO Mesh Group vs 3DMAX Mesh Group; NASA Temporal Demand; Test type: Superiority; p = 0.325, t-test, 1 sided
Statistical Analysis 4: Comparison: ULTRAPRO Mesh Group vs 3DMAX Mesh Group; NASA Peformance; Test type: Superiority; p = 0.0451, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Followed participants for AEs up to 2 years following the procedure.
Description: Evaluation of Surgical Residents Group for All-Cause Mortality, Adverse Events, and Other Adverse Events were not monitored/assessed for Surgical Residents.
Arm/Group | ULTRAPRO Mesh Group | 3DMAX Mesh Group | Evaluation of Surgical Residents
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/0
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-02-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT01825187/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT01825187/ICF_001.pdf